CLINICAL TRIAL: NCT01442025
Title: A Randomized Controlled Trial Investigating Tailored Treatment With Infliximab for Active Luminal Crohn's Disease
Brief Title: Study Investigating Tailored Treatment With Infliximab for Active Crohn's Disease
Acronym: TAILORIX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GETAID 2010-2
Record Dates: First submitted 2011-09-20; First posted 2011-09-28 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; IFX trough level
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 =Control Group (Placebo Comparator): the dose of IFX will be increased by 5 mg/kg (maximally 1 time) based on symptom relapse (usual clinical practice) Dose will be kept stable ofr the rest of the trial Dose decreases will not be allowed.
  Interventions: Drug: Infliximab
- Cohort 2 (Active Comparator): Dose of IFX will be increased by 2.5 mg/kg (maximally 2 times) if the following criteria are met A dose increase is maintained for the following infusions
  Interventions: Drug: Infliximab
- Cohort 3 (Active Comparator): Dose of IFX will be increased by 5 mg/kg (maximally 1 time) if the following criteria are met A dose increase is maintained for the following infusions
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Perfusion of IFX 5mg/kg to be increased to 10 mg/kg based on clinical symptoms
  Other Names: IFX
  Arms: Cohort 1 =Control Group
Drug: Infliximab — Perfusion of IFX 5mg/kg or 10 mg/kg if dose increase criteria are met (biological)
  Other Names: IFX
  Arms: Cohort 2
Drug: Infliximab — Perfusion of IFX 5mg/kg or 7,5 mg/kg if dose increase criteria are met (biological)and 10mg/kg if dose increase criteria are met for a second time
  Other Names: IFX
  Arms: Cohort 3

SUMMARY:
To investigate whether sustained trough levels of IFX can be achieved using IFX (Infliximab) trough level measurements and adjustment of dosing based upon these levels by means of two different standardized algorithms in comparison with 'standard of care' IFX treatment and its effects on clinical and endoscopic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Active CD (CDAI>220) and signs of active inflammation as evidenced by elevated serum hsCRP levels (>5 mg/L) and/or elevated fecal calprotectin levels (>250 µg/g) and endoscopically visible ulcers.
* Patients must be naïve to biologics with indication for starting anti-TNF therapy in accordance with national reimbursement criteria.
* Patients must be naïve to thiopurines or have failed therapy with thiopurines (in which case AZA will be continued).
* Ongoing steroids are allowed if at stable dose for at least 2 weeks and at a maximum of prednisone 40 mg/d or budesonide 9 mg/day.
* Patients who consent to receiving Infliximab 5 mg/kg at week 0, 2 and 6 and further on every 8 weeks in conjunction with azathioprine (2,5 mg/kg/day). Patients who develop AZA intolerance during the trial are continued in the trial without AZA (ie IFX monotherapy).

Exclusion Criteria:

* Absence of endoscopically visible ulcers
* Prior exposure to infliximab (other biologics allowed)
* Ongoing steroid therapy at doses > 40 mg/d prednisolone equivalent
* Previous intolerance to azathioprine leading to drug discontinuation
* Ongoing infections
* Positive tuberculosis screen per local guidelines
* Serious other diseases including cancer in the 5 years prior to inclusion excluding non-melanoma skin cancer
* Indication for immediate surgery
* Pregnant or breast-feeding woman.
* Positive fecal culture for Salmonella, Shigella, Yersinia and Campylobacter and/or presence of Clostridium difficile B toxin in the stools
* Active tuberculosis
* Untreated latent tuberculosis (see national recommendations. Appendix 2).
* Non-compliant subjects.
* Participation in another therapeutic study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Level of remission | 54 weeks after Inclusion
  Proportion of patients with steroid-free remission (CDAI < 150) and endoscopic healing (absence of ulcers) at week 54 CDAI = Crohn's Disease Activity Index

SECONDARY OUTCOMES:
Clinical remission | week 14 after inclusion
  Clinical remission (CDAI <150) at each visit and the whole study period
Endoscopic evaluation | week 0, week 12 and week 54
  * percentage of patients in each group with absence of ulcers;
  * percentage of patients in each group with >50% improvement in CDEIS (Crohn's Disease Endoscopic Index Score

CONTACTS AND LOCATIONS:
Overall Officials: Geert D'Haens, PhD, Study Director — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives; David Laharie, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives
Locations (12):
- France (12):
  - Chu Amiens, Amiens
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - CHRU Lille, Lille
  - CHU NICE, Nice
  - Hopital Saint Louis, Paris
  - CHU Bordeaux - Pessac, Pessac
  - Chu Reims, Reims
  - Chu Rennes, Rennes
  - Chu Toulouse, Toulouse
  - Chu Tours, Tours
  - Chu Nancy, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Hanauer SB, Feagan BG, Lichtenstein GR, Mayer LF, Schreiber S, Colombel JF, Rachmilewitz D, Wolf DC, Olson A, Bao W, Rutgeerts P; ACCENT I Study Group. Maintenance infliximab for Crohn's disease: the ACCENT I randomised trial. Lancet. 2002 May 4;359(9317):1541-9. doi: 10.1016/S0140-6736(02)08512-4. PMID 12047962
- [Background] Sands BE, Anderson FH, Bernstein CN, Chey WY, Feagan BG, Fedorak RN, Kamm MA, Korzenik JR, Lashner BA, Onken JE, Rachmilewitz D, Rutgeerts P, Wild G, Wolf DC, Marsters PA, Travers SB, Blank MA, van Deventer SJ. Infliximab maintenance therapy for fistulizing Crohn's disease. N Engl J Med. 2004 Feb 26;350(9):876-85. doi: 10.1056/NEJMoa030815. PMID 14985485
- [Background] Lemann M, Mary JY, Duclos B, Veyrac M, Dupas JL, Delchier JC, Laharie D, Moreau J, Cadiot G, Picon L, Bourreille A, Sobahni I, Colombel JF; Groupe d'Etude Therapeutique des Affections Inflammatoires du Tube Digestif (GETAID). Infliximab plus azathioprine for steroid-dependent Crohn's disease patients: a randomized placebo-controlled trial. Gastroenterology. 2006 Apr;130(4):1054-61. doi: 10.1053/j.gastro.2006.02.014. PMID 16618399
- [Background] D'Haens G, Baert F, van Assche G, Caenepeel P, Vergauwe P, Tuynman H, De Vos M, van Deventer S, Stitt L, Donner A, Vermeire S, Van De Mierop FJ, Coche JR, van der Woude J, Ochsenkuhn T, van Bodegraven AA, Van Hootegem PP, Lambrecht GL, Mana F, Rutgeerts P, Feagan BG, Hommes D; Belgian Inflammatory Bowel Disease Research Group; North-Holland Gut Club. Early combined immunosuppression or conventional management in patients with newly diagnosed Crohn's disease: an open randomised trial. Lancet. 2008 Feb 23;371(9613):660-667. doi: 10.1016/S0140-6736(08)60304-9. PMID 18295023
- [Background] Baert F, Moortgat L, Van Assche G, Caenepeel P, Vergauwe P, De Vos M, Stokkers P, Hommes D, Rutgeerts P, Vermeire S, D'Haens G; Belgian Inflammatory Bowel Disease Research Group; North-Holland Gut Club. Mucosal healing predicts sustained clinical remission in patients with early-stage Crohn's disease. Gastroenterology. 2010 Feb;138(2):463-8; quiz e10-1. doi: 10.1053/j.gastro.2009.09.056. Epub 2009 Oct 8. PMID 19818785
- [Background] Louis E, Vernier-Massouille G, Grimaud JC, et al. Infliximab discontinuation in Crohn's disease patients in stable remission on combined therapy with immunosuppressors: a prospective ongoing cohort study. Gastroenterology 2009, 136:A-146
- [Background] Rutgeerts P, Diamond RH, Bala M, Olson A, Lichtenstein GR, Bao W, Patel K, Wolf DC, Safdi M, Colombel JF, Lashner B, Hanauer SB. Scheduled maintenance treatment with infliximab is superior to episodic treatment for the healing of mucosal ulceration associated with Crohn's disease. Gastrointest Endosc. 2006 Mar;63(3):433-42; quiz 464. doi: 10.1016/j.gie.2005.08.011. PMID 16500392
- [Background] Colombel JF, Sandborn WJ, Reinisch W, Mantzaris GJ, Kornbluth A, Rachmilewitz D, Lichtiger S, D'Haens G, Diamond RH, Broussard DL, Tang KL, van der Woude CJ, Rutgeerts P; SONIC Study Group. Infliximab, azathioprine, or combination therapy for Crohn's disease. N Engl J Med. 2010 Apr 15;362(15):1383-95. doi: 10.1056/NEJMoa0904492. PMID 20393175
- [Background] Maser EA, Villela R, Silverberg MS, Greenberg GR. Association of trough serum infliximab to clinical outcome after scheduled maintenance treatment for Crohn's disease. Clin Gastroenterol Hepatol. 2006 Oct;4(10):1248-54. doi: 10.1016/j.cgh.2006.06.025. Epub 2006 Aug 22. PMID 16931170
- [Background] Seow CH, Newman A, Irwin SP, Steinhart AH, Silverberg MS, Greenberg GR. Trough serum infliximab: a predictive factor of clinical outcome for infliximab treatment in acute ulcerative colitis. Gut. 2010 Jan;59(1):49-54. doi: 10.1136/gut.2009.183095. PMID 19651627
- [Background] Van Moerkercke W, Ackaert C, Compernolle G, Jürgens M, Cleynen I, Van Assche G, Rutgeerts P, Gils A, Vermeire S. High infliximab trough levels are associated with mucosal healing in Crohn's disease. Gastroenterology 2010; 138 (Supp 1), S-60.
- [Background] Louis E, Collard A, Oger AF, Degroote E, Aboul Nasr El Yafi FA, Belaiche J. Behaviour of Crohn's disease according to the Vienna classification: changing pattern over the course of the disease. Gut. 2001 Dec;49(6):777-82. doi: 10.1136/gut.49.6.777. PMID 11709511
- [Background] Vermeire S, van Assche G, Rutgeerts P. Review article: Altering the natural history of Crohn's disease--evidence for and against current therapies. Aliment Pharmacol Ther. 2007 Jan 1;25(1):3-12. doi: 10.1111/j.1365-2036.2006.03134.x. PMID 17229216
- [Background] Schnitzler F, Fidder H, Ferrante M, Noman M, Arijs I, Van Assche G, Hoffman I, Van Steen K, Vermeire S, Rutgeerts P. Mucosal healing predicts long-term outcome of maintenance therapy with infliximab in Crohn's disease. Inflamm Bowel Dis. 2009 Sep;15(9):1295-301. doi: 10.1002/ibd.20927. PMID 19340881
- [Background] D'haens G, Van Deventer S, Van Hogezand R, Chalmers D, Kothe C, Baert F, Braakman T, Schaible T, Geboes K, Rutgeerts P. Endoscopic and histological healing with infliximab anti-tumor necrosis factor antibodies in Crohn's disease: A European multicenter trial. Gastroenterology. 1999 May;116(5):1029-34. doi: 10.1016/s0016-5085(99)70005-3. PMID 10220494
- [Background] Froslie KF, Jahnsen J, Moum BA, Vatn MH; IBSEN Group. Mucosal healing in inflammatory bowel disease: results from a Norwegian population-based cohort. Gastroenterology. 2007 Aug;133(2):412-22. doi: 10.1053/j.gastro.2007.05.051. Epub 2007 Jun 2. PMID 17681162
- [Background] Rimola J, Rodriguez S, Garcia-Bosch O, Ordas I, Ayala E, Aceituno M, Pellise M, Ayuso C, Ricart E, Donoso L, Panes J. Magnetic resonance for assessment of disease activity and severity in ileocolonic Crohn's disease. Gut. 2009 Aug;58(8):1113-20. doi: 10.1136/gut.2008.167957. Epub 2009 Jan 9. PMID 19136510
- See also: Related Info — http://www.getaid.org